CLINICAL TRIAL: NCT03643458
Title: Splanchnic Oxygenation in Response to Enteral Feeds Before and After Red Blood Cell Transfusion in Preterm Infants
Brief Title: Splanchnic Oxygenation Response to Feeds in Preterm Neonates: Effect of Red Blood Cell Transfusion
Acronym: NIRS_RBC
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-2014-NIRS; 122/2012/U/Oss (Other: Ethic Committee of St.Orsola-Malpighi University Hospital)
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Blood Transfusion Complication; Necrotizing Enterocolitis; Enteral Feeding Intolerance; Preterm Infant
Keywords: NIRS; TANEC; splanchnic oxygenation; enteral feeding; preterm infants
MeSH Terms: conditions — Transfusion Reaction; Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transfused infants: Preterm infants undergone red blood cell transfusion during hospital stay.

SUMMARY:
Since 1987, red blood cell (RBC) transfusions have been proposed as a potential risk factor for necrotizing enterocolitis (NEC), which is one of the most severe gastrointestinal complications of prematurity.

Evidence from Doppler studies have shown a post-transfusion impairment of mesenteric blood flow in response to feeds, whereas NIRS studies have reported transient changes of splanchnic oxygenation after RBC transfusion; a possible role for these findings in increasing the risk for TANEC development has been hypothesized.

The aim of this study is to evaluate SrSO2 patterns in response to enteral feeding before and after transfusion.

DETAILED DESCRIPTION:
Premature neonates are among the most transfused population, but the risks and benefits of this procedure remain unclear. Since 1987, red blood cell (RBC) transfusions have been proposed as a potential risk factor for necrotizing enterocolitis (NEC), which is one of the most common and feared gastrointestinal complications of prematurity. Several observational studies have tried to demonstrate this causal correlation, defining the so-called transfusion-associated NEC (TANEC), which occurs within 48 hours after RBC transfusion.

Evidence from Doppler studies have shown a post-transfusion impairment of mesenteric blood flow in response to feeds, whereas NIRS studies have reported transient changes of splanchnic oxygenation after RBC transfusion. This evidence, which has been hypothesized to play a role on the risk of TANEC development, has significantly raised the attention over the feeding plans during and after RBC transfusion.

To date, splanchnic oxygenation response to feeds before and after transfusion has not been investigated, but could bring useful information to understand the splanchnic hemodynamic changes associated to RBC transfusion.

Therefore, the aim of this study is to evaluate SrSO2 patterns in response to enteral feeding before and after transfusion.

Enrolled infants will undergo a 12-h monitoring of cerebral (CrSO2) and splanchnic (SrSO2) oxygenation, performed using an INVOS 5100 oxymeter (Medtronic, Boulder, CO), whose neonatal sensors will be placed in the central region of the forehead and the below the umbilicus, respectively.

The study monitoring includes the following phases:

* Phase 1 (0-3 hours): pre-transfusion feed and related post-prandial period
* Phase 2 (4-9 hours): RBC transfusion (10 ml/kg),administered over 3 hours, following which feeds are hold for 3 hours.
* Phase 3 (10-12 hours): post-transfusion feed and related post-prandial period.

CrSO2 and SrSO2 patterns before and after transfusion and the related changes from baseline values will be analyzed. SCOR (CrSO2/SrSO2 ratio) patterns will be also calculated and analyzed. IBM SPSS Statistics (Statistical Package for the Social Sciences, SPSS Inc., IBM, Armonk, NY) will be used for statistical analysis. If any infant develops TANEC after transfusion, the related patterns will be evaluated and analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

* gestational age <32 weeks or birth weight <1500 g
* need for red blood cell transfusion according to national guidelines

Exclusion Criteria:

* hemodynamic instability
* Prior occurrence of necrotizing or presence of symptoms and signs of feeding intolerance within one week before transfusion

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Anemic preterm infants requiring red blood cell transfusion.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Pre-transfusion splanchnic oxygenation pattern | Enteral feed before red blood cell transfusion administration (3 hours)
  Decrease or increase of splanchnic oxygenation during and after feed administration compared to pre-prandial baseline value
Post-transfusion splanchnic oxygenation pattern | Enteral feed after red blood cell transfusion administration (3 hours)
  Decrease or increase of splanchnic oxygenation during and after feed administration compared to pre-prandial baseline value

SECONDARY OUTCOMES:
Incidence of gut complications | 48 hours after transfusion
  Occurrence of necrotizing enterocolitis or feeding intolerance in infants undergone red blood cell transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Corvaglia, Principal Investigator — S.Orsola-Malpighi University Hospital, Bologna
Locations (1):
- Neonatal Intensive Care Unit, S.Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marin T, Moore J, Kosmetatos N, Roback JD, Weiss P, Higgins M, McCauley L, Strickland OL, Josephson CD. Red blood cell transfusion-related necrotizing enterocolitis in very-low-birthweight infants: a near-infrared spectroscopy investigation. Transfusion. 2013 Nov;53(11):2650-8. doi: 10.1111/trf.12158. Epub 2013 Mar 11. PMID 23480548
- [Background] White L, Said M, Rais-Bahrami K. Monitoring mesenteric tissue oxygenation with near-infrared spectroscopy during packed red blood cell transfusion in preterm infants. J Neonatal Perinatal Med. 2015;8(2):157-63. doi: 10.3233/NPM-15814090. PMID 26410441
- [Background] Bailey SM, Hendricks-Munoz KD, Mally PV. Variability in splanchnic tissue oxygenation during preterm red blood cell transfusion given for symptomatic anaemia may reveal a potential mechanism of transfusion-related acute gut injury. Blood Transfus. 2015 Jul;13(3):429-34. doi: 10.2450/2015.0212-14. Epub 2015 Jan 30. PMID 25761320
- [Background] Marin T, Josephson CD, Kosmetatos N, Higgins M, Moore JE. Feeding preterm infants during red blood cell transfusion is associated with a decline in postprandial mesenteric oxygenation. J Pediatr. 2014 Sep;165(3):464-71.e1. doi: 10.1016/j.jpeds.2014.05.009. Epub 2014 Jun 16. PMID 24948351
- [Background] Krimmel GA, Baker R, Yanowitz TD. Blood transfusion alters the superior mesenteric artery blood flow velocity response to feeding in premature infants. Am J Perinatol. 2009 Feb;26(2):99-105. doi: 10.1055/s-0028-1090595. Epub 2008 Nov 19. PMID 19021097
- [Background] Banerjee J, Leung TS, Aladangady N. Effect of blood transfusion on intestinal blood flow and oxygenation in extremely preterm infants during first week of life. Transfusion. 2016 Apr;56(4):808-15. doi: 10.1111/trf.13434. Epub 2015 Dec 8. PMID 26643925
- [Background] Banerjee J, Leung TS, Aladangady N. Blood transfusion in preterm infants improves intestinal tissue oxygenation without alteration in blood flow. Vox Sang. 2016 Nov;111(4):399-408. doi: 10.1111/vox.12436. Epub 2016 Aug 10. PMID 27509230